CLINICAL TRIAL: NCT05111834
Title: IRENE-G Study: Impact of Resistance Exercise and Nutritional Endorsement on GvHD Symptoms
Acronym: IRENE-G
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Heidelberg (Other)
Collaborators: Deutsche José Carreras Leukämie-Stiftung (Unknown)
Responsible Party: Principal Investigator, Joachim Wiskemann, Principle Investigator, University Hospital Heidelberg
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: DJCLS 12R/2019
Record Dates: First submitted 2021-09-29; First posted 2021-11-08 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Graft Vs Host Disease
Keywords: Resistance Training; Nutritional Endorsement; Allogenic stem cell transplantation; Steroid-induced myopathy; Cancer; Exercise; Graft versus host disease; Physical performance
MeSH Terms: conditions — Graft vs Host Disease; Neoplasms; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Supervised resistance training plus nutritional endorsement (Experimental): The study participants receive a progressive moderate-to-high-intensity resistance training program (a 60 minutes twice a week for a period of 24- weeks) plus nutritional endorsement. The training will take place at the NCT Heidelberg, in regional qualified facility centers or online under supervision and guidance of experienced exercise therapists.
  The progressive resistance program for participants who train at facility centers comprises of 6 machine-based exercises, each performed 2 sets,12 repetitions of 60%-80% of 1 RM. For participants who train online, the training load will be defined during the introductory training session with the aim of choosing a load which to perform two times 12 repetitions. The program targets major upper and lower body muscle groups (with emphasis on the lower extremities). In addition, patients receive nutritional advice/diet modification, depending on their individual requirements and/or changes in general condition.
  Interventions: Behavioral: Supervised resistance training plus nutritional endorsement
- Nutritional endorsement only (Active Comparator): Patients receive nutritional advice/diet modification, depending on their individual requirements and/or changes in general condition.
  Interventions: Behavioral: Nutritional endorsement

INTERVENTIONS:
Behavioral: Supervised resistance training plus nutritional endorsement — resistance training 2x per week, nutritional endorsement/therapy based on individual needs
  Arms: Supervised resistance training plus nutritional endorsement
Behavioral: Nutritional endorsement — nutritional endorsement/therapy based on individual needs
  Arms: Nutritional endorsement only

SUMMARY:
The IRENE-G trial is a randomized controlled study that aims to investigate the effect of a supervised resistance exercise program (2x/week for 24 weeks) in combination with a nutritional intervention on physical performance/frailty in patients with GvHD symptoms treated with high dose steroids.

DETAILED DESCRIPTION:
Graft-versus-host disease (GvHD) remains the major complication and limitation to successful allogeneic hematopoietic stem cell transplantation (allo-HSCT). Treatment of GvHD is challenging, with high-dose steroids remaining the established first-line treatment in both acute and chronic GvHD. Long-term doses of systemic corticosteroids have many well-known side-effects such as myopathy, though often an overlooked diagnosis. Previous studies in non-cancer patients treated with corticosteroids demonstrated that resistance training can reverse muscle atrophy and weakness. Despite the beneficial effects of exercise, no research effort to date has explicitly examined the effect of a progressive moderate-to-high intensity resistance training on the physical performance and well-being of GvHD patients treated with high-dose steroids. As GvHD patients are commonly found to be malnourished, which affects muscle mass and strength and thus quality of life, nutritional endorsement and optimization should be considered when investigating the effect of exercise in GvHD patients.

The IRENE-G study (acronym for Impact of Resistance Exercise and Nutritional Endorsement on GvHD symptoms) is a 24 week prospective, randomized controlled intervention trial with a two-armed parallel design and 1:1 allocation ratio of GvHD patients treated with high-dose steroids.The exploratory study examines and compares the effects of a supervised resistance exercise intervention - 2x per week, 60 minutes - and a nutritional optimisation program (experimental group) against a nutritional optimisation program only (control group) on physical performance in GvHD patients treated with high-dose steroids. We hypothesize that patients in the experimental group will show significantly greater improvements (or an attenuated decrement) in their physical performance after 24-weeks compared to the control group. Moreover, the investigators hypothesized that the experimental group will have lower levels of fatigue, a higher perceived quality of life, better muscle strength values and a higher vastus lateralis muscle volume, a better nutritional status as well as a better submaximal endurance capacity compared to the control group.

On the basis of power calculations, the goal is to include 56 patients per intervention arm, resulting in a total patient number of n=112.

Assessments will take place at week 8, 16 and 24 after baseline. A follow-up assessment is planned at week 48.

The primary outcome of IRENE-G is physical performance measured via the Short Physical Performance Battery. Further endpoints are muscle strength and volume, submaximal endurance capacity, nutritional status and patient-reported outcomes such as quality of life and fatigue.

ELIGIBILITY:
Inclusion Criteria:

* Existing or new diagnosis of acute or chronic GvHD treated with systemic steroid therapy (≥0,5 mg/kg/day)
* Sufficient German language skills
* Willing/ able to train at the provided exercise facilities or online twice a week
* Willing/ able to take part in the scheduled testing
* Capacity to consent
* Signed informed consent

Exclusion Criteria:

* Any physical or mental conditions that would hamper the adherence to the training and/or nutritional program or the completion of the study procedures
* Heart insufficiency > NYHA III or uncertain arrhythmia
* Uncontrolled hypertension
* Severe renal dysfunction (GFR < 30%, Creatinine> 3mg/dl)
* Reduced standing or walking ability
* Insufficient hematological capacity (either hemoglobin value below 8 g/dl or thrombocytes below 30.000/µL)
* Any other comorbidities that preclude participation in the exercise programs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Estimated)
Dates: Start 2021-09-15 (Actual); Primary Completion 2025-05-31 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Change from baseline to week 24 in Physical performance, as measured by the Short Physical Performance Battery (SPPB) | up to 24 weeks (& 6 month follow-up)
  Physical Performance will be assessed with the Short Physical Performance Battery (SPPB). The SPPB is based on three timed tasks: 4-meter walking speed test, standing balance (feet side-by-side, semi-tandem, full tandem) and sit-to-stand test. Participants score on each component of the battery. Each task is scored out of 4. The sum of the three assessments comprised the final SPPB score with a possible range from 0 to 12. A higher score represents a higher level of function, while lower level indicate lower level of function. Change = (Week 24 Score - Baseline Score). The SPPB is a well-established instrument for the measurement of physical performance, commonly used is elderly patients both in hospital and community setting.

SECONDARY OUTCOMES:
Change from baseline to week 24 in Submaximal endurance performance, assessed with the 6 minute walk test | up to 24 weeks (& 6 month follow-up)
  The 6 minute walk test will be used to determine the submaximal endurance capacity. The test measures the distance an individual is able to walk over a total of six minutes. The goal is for the individual to walk as far as possible within six minutes.
Change from baseline to week 24 in Muscle strength performance, as measured by Hand-held dynamometer | up to week 24 (& 6 month follow-up)
  A hand-held dynamometer will be applied to assess maximal voluntary isometric muscle contraction in Newton meters in 6 muscle groups (knee and elbow flexors and extensors, hip flexors and abductors). Muscle groups will be assessed bilaterally for their isometric power. Change = (Week 24 value - Baseline value)
Change from baseline to week 24 in Muscle volume, assessed with ultrasound measurement | up to week 24 (& 6 month follow-up)
  Ultrasound measurement will be performed to determine the thickness and cross sectional area of both vastus lateralis muscles as well as subcutaneous adipose tissue thickness. Change = (Week 24 value - Baseline value)
Change from baseline to week 24 in Nutritional Status | up to week 24 (& 6 month follow-up)
  The nutritional status will be determined using the Nutritional Risk Screening (NRS 2002), lab parameters (e.g. albumin and total protein), hand-grip strength.
Change from baseline to week 24 Health related Quality of life, as measured by the EORTC QLQ-C30 | up to week 24 (& 6 month follow-up)
  Quality of life will be assessed with the validated 30-item self-assessment questionnaire of the European Organisation for Research and Treatment of Cancer (EORTC QLQ-C30, version 3.0). It comprises five multi-item functional scales (physical, role, emotional, cognitive, and social function), three multi-item symptom scales (fatigue, pain, nausea/vomiting), and six single items assessing further symptoms (dyspnea, insomnia, appetite loss, constipation, diarrhea) and financial difficulties. Scores range from 0 to 100. A higher score for the functional scales and global health status denote a better level of functioning, whereas a high score for symtom/single-item scale indicate a higher level of symptomatology/problems. Change = (Week 24 Score - Baseline Score)
Change from baseline to week 24 in high-dose chemotherapy and stem cell transplantation-related symptoms and problems, as measured by the EORTC QLQ-HDC 29 | up to week 24 (& 6 month follow-up)
  The EORTC QLQ-HDC 29 is a 29-item quality of life questionnaire, which has been developed to elicit patient's experience of symptoms and problems during and after high-dose chemotherapy and stem cell transplantation (57). It consists of 6 multi-item scales (gastro-intestinal side-effects, worry/anxiety, impact on family, body image, sexuality, in-patient issues) and 8 single-item (skin problems, fever/chills, urinary frequency, aches or pain in bones, taking regular drugs, finishing things, ability to have children, experience helping to distinguish what is important in life) questions. Scores range from 0 to 100 with higher score representing higher levels of problems. Change = (Week 24 Score - Baseline Score)
Change from baseline to week 24 in Cancer-related Fatigue, as measured by the EORTC QLQ-FA12 | up to week 24 (& 6 month follow-up)
  Fatigue will be assessed via the EORTC QLQ-FA 12 questionnaire, which is an internationally validated phase IV module of the European Organisation for Research and Treatment of Cancer. The module assesses physical, cognitive and emotional aspects of cancer-related fatigue. It is composed of 12 questions, 10 unidirectional and 2 criteria variables which measure the extent to which fatigue interferes with daily activities and social life. Scores range from 0 to 100. Higher scores represent a higher level of fatigue symptomatology. Change = (Week 24 Score - Baseline Score)
Change from baseline to week 24 in patient-perceived GVHD symptom bother, as measured by the modified 7-day Lee Chronic-versus-Host Disease Symptom Scale | up to week 24 (& 6 month follow-up)
  The modified 7-day Lee Chronic-versus-Host Disease Symptom Scale will be used to capture the GvHD-specific symptom burden. It is a 28 item, 7-domain symptom scale (skin, eyes, mouth, lung, nutrition, energy and psych). Patients will report their level of symptom bother over a period of 7 days on a 5-point Likert scale.
Change from baseline to week 24 in Functional Status determined with the Karnofsky performance scale | up to week 24 (& 6 month follow-up)
  The Karnofsky performance scale (KPS) will be applied to assess functional status of a patient. The KPS is a 11-point rating scale, which ranges from normal functioning (100%) to dead (0%). The scale is widely used due to its psychometric properties and recommended in clinical assessments.

CONTACTS AND LOCATIONS:
Overall Officials: Joachim Wiskemann, PD Dr., Principal Investigator — Heidelberg University Hospital, National center for Tumor Diseases, Division of Medical Oncology
Locations (1):
- Heidelberg University Hospital, Heidelberg, Germany, Germany

REFERENCES:
- [Derived] Ernst M, Wagner C, Oeser A, Messer S, Wender A, Cryns N, Brockelmann PJ, Holtkamp U, Baumann FT, Wiskemann J, Monsef I, Scherer RW, Mishra SI, Skoetz N. Resistance training for fatigue in people with cancer. Cochrane Database Syst Rev. 2024 Nov 28;11(11):CD015518. doi: 10.1002/14651858.CD015518. PMID 39606939
- [Derived] Bujan Rivera J, Kuhl R, Zech U, Hendricks A, Luft T, Dreger P, Friedmann-Bette B, Betz TM, Wiskemann J. Impact of Resistance Exercise and Nutritional Endorsement on physical performance in patients with GvHD (IRENE-G study) - design and rational of a randomized controlled trial. BMC Cancer. 2022 Apr 22;22(1):440. doi: 10.1186/s12885-022-09497-1. PMID 35459108